CLINICAL TRIAL: NCT01917838
Title: Mobile Health Solutions for Behavioral Skill Implementation Through Homework
Acronym: MHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Silver School of Social Work (Other)
Responsible Party: Principal Investigator, Mary M. McKay, McSilver Professor of Poverty Studies, Director, McSilver Institute for Poverty Policy and Research, NYU Silver School of Social Work
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R34MH100407-01 (NIH)
Record Dates: First submitted 2013-07-18; First posted 2013-08-07 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Mental Health Wellness 1
Keywords: Mental Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MFG plus MyMFG (Experimental): MFG plus MyMFG will be tested and the aim is:
  1. Greater quality of the "Design" and "Do" process rated by therapists, parents, and independent coders.
  2. Greater quantity and quality of HW assignments rated by therapists and parents.
  3. Greater quality of the "Review" process as rated by therapists, parents, and independent coders.
  4. Greater satisfaction with treatment as rated by the parent, target child, and therapists.
  Interventions: Behavioral: MFG plus MyMFG

INTERVENTIONS:
Behavioral: MFG plus MyMFG — Specific aim is to utilize mHealth to improve the "Design" and "Do" process of HW within the context of the Family Groups for Youth with Behavioral Difficulties (MFG) intervention, an EBT for DBDs in youth and their families who seek assistance at outpatient mental health clinics in urban communities.
  The first component focuses on delivering HW via a highly engaging, multiplayer, interactive, cooperative, and skill-building game platform aimed at improving the "Design" and "Do" process of HW. The second component focuses on targeting factors putatively related to poor HW implementation within the "Do" process.

SUMMARY:
The goal of this two-year R34 treatment development grant is to develop a mobile health (mHealth) application that will both advance theory in and clinical practice of homework (HW) implementation.

HW can be described as between-session exercises where the client practices specific skills learned within-session in order to promote skill acquisition, which ultimately leads to improved acute- as well as longer-term therapeutic benefits on targeted outcomes, generalization of treatment effects and maintenance of treatment gains. Despite data demonstrating that HW is critical to achieving maximal benefits from evidence-based treatments, very little theory-driven approaches have been conducted focusing on improving the HW process. Through utilizing self-determination theory as a guiding framework and integrating principles from the field of "gamification" and goal-setting, the aim is to develop a two-component mHealth HW application (My MFG).

The first component focuses on delivering HW via a highly engaging, multiplayer, interactive, cooperative, and skill-building game platform aimed at improving the "Design" and "Do" process of HW. The second component focuses on targeting factors putatively related to poor HW implementation within the "Do" process.

The process of the development of My MFG will be guided by the clinic and community development model and iterative software development process to maximize the feasibility and sustainability of My MFG within practice settings often characterized by limited resources. Findings from this study have broad implications for evidence-based treatments for youth and adult mental health disorders that emphasize HW as the link between treatment and improvements in targeted outcomes.

DETAILED DESCRIPTION:
The aim of the proposed study is to develop a theory-informed mobile health (mHealth) application for urban caregivers attempting to improve their children's oppositional and conduct related difficulties (i.e., disruptive behavior disorders; DBDs). The majority of evidence-based treatments (EBTs) targeting youth DBDs emphasize change in specific parenting/family-level processes empirically linked to the maintenance of DBDs. Existing EBTs frequently include at-home-practice-exercises (i.e., homework; HW) to reinforce parent skill acquisition and maximize use of new skills with children at home. Poor quantity and quality of HW completed by parents significantly attenuates the effect of EBTs. This is a significant limiting-factor in many EBTs attaining full public health impact. Given the robust effect of HW on outcomes from EBTs across a range of behavioral health difficulties and populations, there is a call for moving beyond the question of whether HW is important to questions such as what processes are involved in HW implementation and how best to support these processes. Minimal investigation has been focused on these critical questions.

A model of HW has recently been proposed to better understand the process of HW implementation, as well as guide critically needed supports for at-home practice exercises.

This model proposes four HW processes:

1. Designing;
2. Assigning;
3. Doing, and;
4. Reviewing.

The DADR model proposes that specific social, cognitive and behavioral factors related to the HW task, as well as to the provider and the adult caregiver may affect the quality of each phase and ultimately to the quantity and quality of HW completed. Methods to better understand, support, and impact these processes are essential to advancing theory and offering solutions to HW completion.

Through features available on smartphones (e.g., camera/video/voice recording; simple message service; internet-access; global positioning system), there are novel methods to interface with and support clients outside of defined treatment sessions. Through the use of these features, mHealth applications can be used to engage, educate, connect, track, and remind clients. These applications can use push (send communications) or pull (client's access tools on their own) mechanisms to engage the client in behavioral change activity. mHealth applications that integrate push and pull methods offer a significant opportunity to enhance outcomes across a range of health and behavioral health challenges and populations.

The goal of this two-year R34 treatment development grant is in response to RFA-MH-13-061 (Harnessing advanced health technologies to drive mental health improvement) to develop a mHealth application that will both advance theory in and clinical practice guided by the DADR model of HW implementation. Specifically we aim to utilize mHealth to improve the "Design" and "Do" process of HW within the context of the Family Groups for Youth with Behavioral Difficulties (MFG) intervention, an EBT for DBDs in youth and their families who seek assistance at outpatient mental health clinics in urban communities. To date, efforts at utilizing mHealth within the context of HW have been minimal and have not taken a systematic, theory-driven approach, thereby limiting the advance of knowledge and clinical application. Through utilizing self-determination theory as a guiding framework and integrating principles from the field of "gamification" and goal-setting, the aim is to develop a two-component MFG mHealth HW application (My MFG). The first component focuses on delivering MFG HW via a highly engaging, multiplayer, interactive, cooperative, and skill-building game platform aimed at improving the "Design" and "Do" process. The second component focuses on targeting factors putatively related to poor HW implementation within the "Do" process.

The process of the development of My MFG will be guided by the clinic and community development model and iterative software development process to maximize the feasibility and sustainability of My MFG within practice settings often characterized by limited resources. The specific aims of this project are to:

1. Develop My MFG through an iterative process informed by the perspectives of key stakeholders
2. Determine the impact of MFG plus My MFG relative to MFG-alone on the DADR process and HW quantity and quality. It is hypothesized that the MFG plus My MFG will result in:

   1. Greater quality of the "Design" and "Do" process rated by therapists, parents, and independent coders
   2. Greater quantity and quality of HW assignments rated by therapists and parents
   3. Greater quality of the "Review" process as rated by therapists, parents, and independent coders as a function of improved HW quantity and quality
   4. Greater satisfaction with treatment as rated by the parent, target child, and therapists NIMH has specifically called for acceleration of research to maximize the ability of current treatments to reduce symptoms, improve adherence and functioning while improving quality of and lowering the cost of care. The mHealth application and methods proposed herein serve as systematic, theory-driven approaches to significantly advance understanding of how best to support the HW process-a common element of many EBTs across various disorders and populations-ultimately resulting in greater effectiveness of EBTs, maintenance and generalization of behavioral skills learned during EBTs.

ELIGIBILITY:
Inclusion Criteria:

1) youth between the ages of 7 to 13 years and an accompanying adult primary caregiver available to participate in the research and intervention activities 2) English speaking youth and adult caregiver and 3) youth meeting criteria for DBD via parent reports based on the Disruptive Behavior Disorder (DBD) rating scales of DSM symptoms and cross-situational impairment as assessed through parent ratings on the Impairment Rating Scale (IRS). Children will be diagnosed with DBD if they meet DSM symptom criteria for DBD by parent report (i.e., at least four symptoms of ODD or 3 symptoms of CD), and impairment ratings indicate at least one impairment domain.

-

Exclusion Criteria:

Children will also be excluded if there is:

* Evidence of psychosis
* If the youth or adult caregiver presents with emergency psychiatric needs that require services beyond that which can be managed within an outpatient setting (e.g. hospitalization, specialized placement outside the home), active intervention by clinic and research staff to secure what is needed will be made
* Children will not be excluded if they participate in other psychosocial or pharmacological interventions.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
DADR Process- HW quantity and quality, Homework Rating Scale-II | Weekly for 16 weeks; duration of group
  This assessment helps to understand the DADR process and to assess if homework was completed and how much.
DADR Proces- Homework Adherence and Competence Scales | Participants will be tracked up to 16 weeks and feedback will be collected every week.
  An independent observer will assess level of homework adherence and competence in every session.

SECONDARY OUTCOMES:
DBD Symptoms -DBD Rating Scale | Day 1- 1st contact
  To assess the severity of behavior problems.
Children's Impairment Rating Scale | Day 1- 1st Contact
  To assess level of behavioral impairment for child- caregiver reports.
Attendance | Weekly- duration of the 16 week group
  Attendance will be measured for each participant at every session.
IOWA Conners Oppositional/Defiant Scale | 1st contact and at the end of the 16 week group
  Caregiver assesses child's oppostitional and defiant behaviors at pre and post treatment.
Consumer Satisfaction & Feedback- Treatment Attitude Inventory | 1st contact and at the end of the 16 week group
  This is a feedback assesment that will happen at either group or individual consultancy meeting to assess feedback of the MHealth process by parent, target child, and therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Mary M McKay, PhD, Principal Investigator — New York University Silver School of Social Work; Tyrone M Parchment, LMSW, Study Director — New York University Silver School of Social Work; Ozge Sensoy-Bahar, PhD, Study Director — New York University Silver School of Social Work
Locations (1):
- McSilver Institute for Poverty Policy and Research - New York University Silver School of Social Work, New York, New York, United States

REFERENCES:
- [Derived] Chacko A, Isham A, Cleek AF, McKay MM. Using mobile health technology to improve behavioral skill implementation through homework in evidence-based parenting intervention for disruptive behavior disorders in youth: study protocol for intervention development and evaluation. Pilot Feasibility Stud. 2016 Sep 20;2:57. doi: 10.1186/s40814-016-0097-4. eCollection 2016. PMID 27965873